CLINICAL TRIAL: NCT07319195
Title: Window of Opportunity Study of Intratumoral CD40 Agonist (Mitazalimab) With or Without PD-1 Inhibitor (Nivolumab) in Patients With Resectable Breast Cancer (WINIT-BC)
Brief Title: Window Study of Intratumoral Mitazalimab in Breast Cancer (WINIT-BC)
Acronym: WINIT-BC
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jennifer Zhang (Other)
Collaborators: Alligator Bioscience AB (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Zhang, Assistant Professor of Surgery at the Hospital of the University of Pennsylvania, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 858844
Record Dates: First submitted 2025-11-26; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: resectable breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (DL-1) (Experimental): Arm A: Intratumoral Mitazalimab 22.5 ug/kg. This dose level will only be explored if ≥ 2 DLTs occur at any time in DL1.
  Interventions: Drug: Intratumoral Mitazalimab
- Arm A (DL 0) (Experimental): Intratumoral Mitazalimab 75 ug/kg
  Interventions: Drug: Intratumoral Mitazalimab
- Arm A (DL+1) (Experimental): Intratumoral Mitazalimab 200 ug/kg
  Interventions: Drug: Intratumoral Mitazalimab
- Arm B (DL-1) (Experimental): Intratumoral Mitazalimab 22.5 ug/kg + intratumoral Nivolumab This dose level will only be explored if ≥ 2 DLTs occur at any time in DL1.
  Interventions: Drug: Intratumoral Mitazalimab; Drug: Intratumoral Nivolumab
- Arm B (DL 0) (Experimental): Intratumoral Mitazalimab 75 ug/kg + intratumoral Nivolumab
  Interventions: Drug: Intratumoral Mitazalimab; Drug: Intratumoral Nivolumab
- Arm B (DL+1) (Experimental): Intratumoral Mitazalimab 200 ug/kg + intratumoral Nivolumab
  Interventions: Drug: Intratumoral Mitazalimab; Drug: Intratumoral Nivolumab

INTERVENTIONS:
Drug: Intratumoral Mitazalimab — Intratumoral agonistic CD40
Drug: Intratumoral Nivolumab — Checkpoint inhibitor
  Arms: Arm B (DL 0); Arm B (DL+1); Arm B (DL-1)

SUMMARY:
The goal of this clinical trial is to study the safety, feasibility, histologic and immunological effects of Mitazalimab, a CD40 agonistic antibody, when administered either alone or in combination with PD-1 inhibition prior to surgical resection.

The investigator hypothesizes that preoperative administration of CD40 agonist with or without PD-1 inhibitor intratumorally will demonstrate an acceptable safety profile, will not result in an unplanned delay in surgery, and will lead to increased immune activation.

Subjects will receive a single intratumoral dose of CD40 agonist with or without PD-1 inhibitor 7 or more days prior to surgery and will be followed for safety, feasibility, immune, and pathologic responses.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written IRB-approved informed consent.
2. Age ≥18 years.
3. Body weight > 30kg
4. Stage I-III or recurrent resectable breast cancer to be treated with curative-intent
5. Planning to undergo upfront surgery as part of routine clinical care
6. Discussion with the treating or study medical oncologist re: the potential of sending an Oncotype evaluation (if ER+HER2-) on the core needle biopsy sample
7. Availability of the core needle biopsy sample for correlative studies
8. Surgery to be performed at a University of Pennsylvania Hospital
9. Life expectancy of at least 12 weeks.
10. Adequate bone marrow, hepatic, and renal function. ANC (Absolute Neutrophil Count) ≥ 1.5x109 cell/ml, platelets ≥75,000 /mm3, hemoglobin ≥9.0 g/dL, total serum bilirubin within 1.5 x upper limit of normal (ULN) unless Gilbert's, AST/ALT, within 2.5 x ULN, Albumin ≥3g/dL, and all tests performed within 4 weeks prior to administration of Study Treatment.
11. ECG with no clinically significant findings as assessed by the investigator.
12. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1.
13. Female patients of childbearing potential who are not abstinent and intend to be sexually active with a non-sterilized male partner must use at least 1 highly effective method of contraception from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after therapy). Non-sterilized male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period. Female patients should also refrain from breastfeeding throughout this period.
14. Able and willing to comply with all study procedures.

Exclusion Criteria:

1. Metastatic disease.
2. Planned neoadjuvant therapy, i.e., not undergoing upfront surgery.
3. Known history of hepatitis B or C with active viral replication.
4. Administration of any live vaccine within 28 days of first dose of study treatment.
5. Prior CD40 or anti-PD-1 agonist therapy.
6. Participation in another interventional clinical trial within 30 days before receiving first dose of study treatment. However, the subject may participate in observational studies.
7. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.
8. Current or prior use of immunosuppressive medication within 14 days before study treatment. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
9. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
10. History of allogenic organ transplantation
11. Active or prior documented autoimmune disease. Examples include inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]. The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or type 1 DM controlled with insulin
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active autoimmune disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
12. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
13. History of another active malignancy except for non-melanoma skin cancer, lentigo maligna or other carcinoma in situ
14. History of active primary immunodeficiency
15. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
16. Body weight > 110 kg.
17. Actively breastfeeding. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 3 or higher adverse events as assessed by CTCAE v5.0 | Within 30 days of treatment
  Type and severity of adverse events
Feasibility of CD40 agonist (Mitazalimab) with/without PD-1 inhibitor (Nivolumab) prior to surgery | 14 days after planned surgical date
  Number of successful surgical resection without unanticipated delay in surgery > 14 days after planned surgical date due to treatment-related issues

SECONDARY OUTCOMES:
Tumor response rate | 2 weeks after surgery
  Rate of tumors with response (Residual Cancer Burden 0-II)
Recurrence of disease | up to 5 years post surgery
  Occurrence of a breast cancer recurrence
Event-free survival | up to 5 years post surgery
  Length of time between time of surgery and a breast cancer recurrence or death
immunologic effects of CD40 agonist (Mitazalimab) with/without PD-1 inhibitor (Nivolumab) | Prior to treatment and up to 30 days post surgery
  Immunophenotyping of PBMCs pre- and post-treatment
Number of participants with change in serum cytokine levels pre- and post-treatment | Prior to treatment and up to 30 days post surgery
  Serum cytokine measurement
Number of participants with changes in tumor immune cell number pre- and post-treatment | Prior to treatment and up to 30 days post surgery
  10x genomics platform will be used to evaluate for changes in tumor immune cell number pre- and post-treatment
Number of participants with changes in TCR repertoire in peripheral blood pre- and post-treatment | Prior to treatment and up to 30 days post surgery
  Comparison of TCR repertoire in peripheral blood via TCR sequencing pre- and post-treatment
Number of participants with changes in TCR repertoire in tumor pre- and post-treatment | Prior to treatment and up to 30 days post surgery
  Comparison of TCR repertoire in tumor via TCR sequencing pre- and post-treatment
Number of patients with FDG PET/CT response or flair after treatment | between baseline and 1 week post-treatment
  Change in FDG activity in tumor and/or lymph nodes between baseline (PET0) and post-treatment (PET1) FDG PET/CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Zhang, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No